CLINICAL TRIAL: NCT01074879
Title: Effects of Protein Quantity and Quality in Combination With Resistance Exercise on Muscle Mass and -Strength in Icelandic Elderly.
Brief Title: Protein Ingestion and Resistance Exercise in Elderly
Acronym: IceProQualita
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iceland (Other)
Collaborators: Landspitali University Hospital Research Fund (Other)
Responsible Party: Prof. Inga Thorsdottir
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 071323007
Record Dates: First submitted 2010-02-23; First posted 2010-02-24 (Estimated); Last update posted 2010-02-24 (Estimated); Status verified 2010-02

CONDITIONS: Healthy
Keywords: Elderly; protein consumption; resistance exercise; muscle mass
MeSH Terms: interventions — Whey Proteins; Milk Proteins; Carbohydrates

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Whey protein (Experimental): 20 g whey protein + 20 g carbohydrates
  Interventions: Dietary Supplement: Whey protein
- Milk protein (Experimental): 20 g milk protein + 20 g carbohydrates
  Interventions: Dietary Supplement: Milk protein
- Carbohydrates (Active Comparator): 40 g carbohydrates
  Interventions: Dietary Supplement: Carbohydrates

INTERVENTIONS:
Dietary Supplement: Whey protein — Dietary supplement after training
  Arms: Whey protein
Dietary Supplement: Milk protein — Dietary supplement after training
  Arms: Milk protein
Dietary Supplement: Carbohydrates — Dietary supplement after training
  Arms: Carbohydrates

SUMMARY:
The mail goal of this randomized controlled, dietary intervention study is to investigate whether protein supplementation in combination with resistance exercise can increase muscle mass and strength in elderly. Loss of muscle mass and -strength is frequent in this group. Participants (N = 220, equal distribution between men and women) are randomized to one of three groups receiving different quantities and qualities of protein supplementation after exercise. The results of this study will be used to form recommendations regarding diet and exercise for the prevention of this frequent health problem in elderly.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and older

Exclusion Criteria:

* uncontrolled coronary heart disease
* pharmacological interventions with drugs known to affect muscle mass
* major orthopedic disease
* low cognitive function.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 220 (Actual)
Dates: Start 2008-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Unit for Nutrition Research, Reykjavik, Iceland

REFERENCES:
- [Derived] Og G, M C, Pv J, I T, A R. Associations of physical activity with vitamin D status depends on obesity status in old adults. Clin Nutr ESPEN. 2020 Oct;39:222-226. doi: 10.1016/j.clnesp.2020.06.009. Epub 2020 Jul 12. PMID 32859321
- [Derived] Geirsdottir OG, Chang M, Jonsson PV, Thorsdottir I, Ramel A. Obesity, Physical Function, and Training Success in Community-Dwelling Nonsarcopenic Old Adults. J Aging Res. 2019 Feb 18;2019:5340328. doi: 10.1155/2019/5340328. eCollection 2019. PMID 30906596
- [Derived] Geirsdottir OG, Chang M, Briem K, Jonsson PV, Thorsdottir I, Ramel A. Gender, Success, and Drop-Out during a Resistance Exercise Program in Community Dwelling Old Adults. J Aging Res. 2017;2017:5841083. doi: 10.1155/2017/5841083. Epub 2017 Aug 14. PMID 28890833
- [Derived] Arnarson A, Gudny Geirsdottir O, Ramel A, Jonsson PV, Thorsdottir I. Insulin-Like Growth Factor-1 and Resistance Exercise in Community Dwelling Old Adults. J Nutr Health Aging. 2015 Oct;19(8):856-60. doi: 10.1007/s12603-015-0547-3. PMID 26412290
- [Derived] Ramel A, Geirsdottir OG, Jonsson PV, Thorsdottiri I. C-Reactive Protein and Resistance Exercise in Community Dwelling Old Adults. J Nutr Health Aging. 2015 Aug;19(7):792-6. doi: 10.1007/s12603-015-0548-2. PMID 26193865
- [Derived] Geirsdottir OG, Arnarson A, Ramel A, Briem K, Jonsson PV, Thorsdottir I. Muscular strength and physical function in elderly adults 6-18 months after a 12-week resistance exercise program. Scand J Public Health. 2015 Feb;43(1):76-82. doi: 10.1177/1403494814560842. Epub 2014 Nov 27. PMID 25431460
- [Derived] Arnarson A, Ramel A, Geirsdottir OG, Jonsson PV, Thorsdottir I. Changes in body composition and use of blood cholesterol lowering drugs predict changes in blood lipids during 12 weeks of resistance exercise training in old adults. Aging Clin Exp Res. 2014 Jun;26(3):287-92. doi: 10.1007/s40520-013-0172-0. Epub 2013 Dec 1. PMID 24293371
- [Derived] Geirsdottir OG, Arnarson A, Ramel A, Jonsson PV, Thorsdottir I. Dietary protein intake is associated with lean body mass in community-dwelling older adults. Nutr Res. 2013 Aug;33(8):608-12. doi: 10.1016/j.nutres.2013.05.014. Epub 2013 Jun 27. PMID 23890349
- [Derived] Arnarson A, Gudny Geirsdottir O, Ramel A, Briem K, Jonsson PV, Thorsdottir I. Effects of whey proteins and carbohydrates on the efficacy of resistance training in elderly people: double blind, randomised controlled trial. Eur J Clin Nutr. 2013 Aug;67(8):821-6. doi: 10.1038/ejcn.2013.40. Epub 2013 Mar 13. PMID 23486511
- [Derived] Ramel A, Arnarson A, Geirsdottir OG, Jonsson PV, Thorsdottir I. Glomerular filtration rate after a 12-wk resistance exercise program with post-exercise protein ingestion in community dwelling elderly. Nutrition. 2013 May;29(5):719-23. doi: 10.1016/j.nut.2012.10.002. Epub 2013 Jan 11. PMID 23317926
- [Derived] Geirsdottir OG, Arnarson A, Briem K, Ramel A, Jonsson PV, Thorsdottir I. Effect of 12-week resistance exercise program on body composition, muscle strength, physical function, and glucose metabolism in healthy, insulin-resistant, and diabetic elderly Icelanders. J Gerontol A Biol Sci Med Sci. 2012 Nov;67(11):1259-65. doi: 10.1093/gerona/gls096. Epub 2012 Apr 10. PMID 22496538
- [Derived] Geirsdottir OG, Arnarson A, Briem K, Ramel A, Tomasson K, Jonsson PV, Thorsdottir I. Physical function predicts improvement in quality of life in elderly Icelanders after 12 weeks of resistance exercise. J Nutr Health Aging. 2012 Jan;16(1):62-6. doi: 10.1007/s12603-011-0076-7. PMID 22238003